CLINICAL TRIAL: NCT01321450
Title: Economisation of Preparation by Using an Ultrasonic Dissection Device in Partial Pancreatoduodenectomy
Brief Title: Economisation of Whipple Resection Using an Ultrasonic Dissection Device
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2908
Record Dates: First submitted 2011-01-24; First posted 2011-03-23 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Resectable Pancreatic Head Neoplasm; Resectable Periampullary Neoplasm; Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Preparation with Harmonic WAVE
- Group B: Preparation with conventional modalities

SUMMARY:
Including 150 randomised patient, the studies aim is to determine whether an economisation and/or improvement in terms of operating time, drainage fluid, blood loss, time of hospitalisation can be found using an ultrasonic dissection device versus traditional surgical methods such as stitches an ligations.The study is performed for patients undergoing partial pancreatoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

resectable tumor

Exclusion Criteria:

palliative resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for partial pancreatoduodenectomy for pancreatic head carcinoma, periampullary carcinoma, chronic pancreatitis and other benign lesions.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Total operation time | end of operation
  Measurement of time regarding incision-closure-time

SECONDARY OUTCOMES:
intraoperative blood loss | end of operation
number of transfusions | within the first 24 hours perioperatively
hospitalization time | end of hospitalization
resulting cost reduction | end of hospitalization
pancreatic fistula | within the first 5 days postoperatively
postoperative intervention | end of hospitalization
  Postoperative interventions due complications, e.g. pancreatic fistula

CONTACTS AND LOCATIONS:
Overall Officials: Jacob R. Izbicki, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (3):
- UH Eppendorf, Hamburg, Germany
- Agia Olga hospital, Athens, Greece
- UH Verona, Verona, Italy

REFERENCES:
- [Background] Ujiki MB, Talamonti MS. Guidelines for the surgical management of pancreatic adenocarcinoma. Semin Oncol. 2007 Aug;34(4):311-20. doi: 10.1053/j.seminoncol.2007.05.004. PMID 17674959
- [Background] Hruby GW, Marruffo FC, Durak E, Collins SM, Pierorazio P, Humphrey PA, Mansukhani MM, Landman J. Evaluation of surgical energy devices for vessel sealing and peripheral energy spread in a porcine model. J Urol. 2007 Dec;178(6):2689-93. doi: 10.1016/j.juro.2007.07.121. Epub 2007 Oct 22. PMID 17945280
- [Background] Nicastri DG, Wu M, Yun J, Swanson SJ. Evaluation of efficacy of an ultrasonic scalpel for pulmonary vascular ligation in an animal model. J Thorac Cardiovasc Surg. 2007 Jul;134(1):160-4. doi: 10.1016/j.jtcvs.2007.02.015. PMID 17599502
- [Derived] Uzunoglu FG, Stehr A, Fink JA, Vettorazzi E, Koenig A, Gawad KA, Vashist YK, Kutup A, Mann O, Gavazzi F, Zerbi A, Bassi C, Dervenis C, Montorsi M, Bockhorn M, Izbicki JR. Ultrasonic dissection versus conventional dissection techniques in pancreatic surgery: a randomized multicentre study. Ann Surg. 2012 Nov;256(5):675-9; discussion 679-80. doi: 10.1097/SLA.0b013e318271cefa. PMID 23095609
- See also: UH Hamburg-Eppendorf - General, Visceral and Thoracic Surgery Department and Clinic — http://www.uke.de/kliniken/allgemeinchirurgie/